CLINICAL TRIAL: NCT02577861
Title: Multinational, Multicentre, Prospective, Open-label, Uncontrolled Clinical Trial to Assess the Efficacy and Safety of Autologous Cultivated Limbal Stem Cells Transplantation (ACLSCT) for Restoration of Corneal Epithelium in Patients With Limbal Stem Cell Deficiency Due to Ocular Burns (HOLOCORE)
Brief Title: Efficacy and Safety of Autologous Cultivated Limbal Stem Cells Transplantation (ACLSCT) for Restoration of Corneal Epithelium in Patients With Limbal Stem Cell Deficiency
Acronym: HOLOCORE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Holostem s.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCD-GPLSCD01-03; 2014-002845-23 (EudraCT Number)
Record Dates: First submitted 2015-10-15; First posted 2015-10-16 (Estimated); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Limbal Stem Cells Deficiency
Keywords: limbal stem cells deficinecy, LSCD, ocular burn
MeSH Terms: interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Holoclar (Experimental): Treatment with Holoclar (medicinal product), including biopsy, graft production and implantation of the graft containing stem cell
  Interventions: Procedure: Biopsy from donor eye; Procedure: Implant of Holoclar; Procedure: Ophtalmologic examination; Procedure: Blood sample collection; Procedure: Digital pictures; Procedure: ECG; Behavioral: Questionnaires; Procedure: Physical examination and vital signs

INTERVENTIONS:
Procedure: Biopsy from donor eye — Corneal biopsy from undamaged limbus
Procedure: Implant of Holoclar — Implant of Holoclar into the eye to be treated after scraping of the fibrovascular pannus
  Other Names: ACLSCT
Procedure: Ophtalmologic examination — The following assessments are performed:
  Epithelial defects assessment by fluorescein staining; superficial corneal neo-vascularization assessment; Best-Corrected Visual Acuity; ocular tonometry; slit lamp examination (both corneal endothelium and anterior chamber); conjunctival inflammation (both bulbar and limbal) assessment; corneal sensitivity and involvement assessment; Schirmer's test type I; evaluation of the following symptoms: pain, burning, photophobia.
Procedure: Blood sample collection — Standard haematology, biochemistry and Infectious profile (Virology) are assessed
Procedure: Digital pictures — At least 4 digital corneal slit lamp photos without fluorescein and at least 4 digital corneal slit lamp photos with fluorescein are taken using digital camera
Procedure: ECG — A 12-lead ECG measurement in single recording at screening for safety reason and before each transplantation.
Behavioral: Questionnaires — Quality of Life assessment through the NEI VFQ 25and EQ-5D-3L questionnaire (EQ-5D-Y in paediatric population)
Procedure: Physical examination and vital signs — A complete physical examination and vital signs (Systolic and Diastolic Blood Pressure (SBP, DBP) and Pulse Rate (PR) must be assessed at each visit (but not at pre-screening and at visit 6)

SUMMARY:
The purpose of this trial is to confirm the efficacy of Holoclar at one year after the first treatment in patients suffering from moderate to severe LSCD (Limbal Stem Cell Deficiency) secondary to ocular burns. In case of failure of the treatment and upon clinical indication of the Principal Investigator, a second transplant with Holoclar will be offered if eligibility will be confirmed. The efficacy of two treatments with Holoclar at one year after the last treatment will be also evaluated. All patients will be followed-up for 12 months after each implant to determine the treatment efficacy by an Independent Assessor.

DETAILED DESCRIPTION:
This is a multinational, multicentre, prospective, open label, uncontrolled clinical trial.

Patients will be screened according to the Study Inclusion and Exclusion criteria and will be candidates for the ACLSCT if all eligibility criteria are met.

Patients then will undergo limbal biopsy for the collection of limbal stem cells for product manufacturing. The confirmation of the eligibility criteria is followed by a roll-in phase of approximately 6 months. At the end of the roll-in period, Holoclar will be implanted through a specific surgical procedure.

After ACLSCT, efficacy assessments will be performed at 1, 3, 6, 9 and 12 months for both first and second treatment (the latter only when applicable). One year after the transplantation, efficacy will be adjudicated by two independent assessors (primary and key secondary endpoints) and the study completion will be reached when 1 year of follow-up after the last transplant in the last patient will be accomplished.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to any study-related procedures.
2. Adult male and female patients (≥18 years old); Five Paediatric patients aged 2 to 17 years will be also enrolled for safety purposes only.
3. LSCD secondary to unilateral or bilateral physical or chemical ocular burns, with at least 1-2 mm2 of undamaged limbus to harvest stem cells for expansion in culture. LSCD will be considered for inclusion in presence of superficial neo-vascularization invading at least two corneal quadrants with central corneal involvement (including corneal neo-vascularisation, corneal opacity or corneal dyschromia) according to the independent assessors;
4. Stability of LSCD, defined by a duration of disease of at least 24 months at the time of the Screening Visit and presence of continuum epithelium as per fluorescein staining scored as none or trace.
5. Presence of severe impairment in visual acuity defined by a score of 1/10th or below 20/200 at the Snellen chart (legal blindness) after best correction (i.e. Best Corrected Visual Acuity);
6. Absence of other clinical contraindications to ACLSC transplantation based upon investigator's judgment;
7. A cooperative attitude to follow up the study procedures (Caregivers in case of minors).

Exclusion Criteria:

1. LSCD of mild degree (i.e. below 2 quadrants of neo-vessel invasion without central corneal), due to a recent burn (less than 24 months before screening), or secondary to medical conditions other than burns (i.e. radiotherapy);
2. Severe ocular inflammation according to the Efron Grading Scale for Contact Lens Complications. Patient can be re-screened after appropriate treatment;
3. Presence of eyelids malposition;
4. Conjunctival scarring with fornix shortening;
5. Severe tear secretion deficiency, determined by Schirmer's test type I (<5 mm/ 5 min);
6. Corneal anaesthesia and conjunctival anaesthesia;
7. Active local or systemic infections at the time of screening. Patient can be re-screened after appropriate treatment;
8. Diagnosis of local or systemic neoplastic disease;
9. Congenital diseases (i.e., Aniridia);
10. Bilateral inflammatory diseases (i.e. Stevens-Johnson syndrome, phemphigoid);
11. A pre-existing blindness precluding a functional recovery;
12. Female subjects: pregnant or lactating women and all women physiologically capable of becoming pregnant (i.e. women of childbearing potential) UNLESS are willing to use one or more reliable methods of contraception (i.e. contraceptive methods other than oral contraceptives, IUD, tubal ligature). Reliable contraception should be maintained throughout the study. Any postmenopausal women (physiologic menopause defined as "12 consecutive months of amenorrhea") or women permanently sterilized (e.g. tubal occlusion, hysterectomy or bilateral salpingectomy) may be enrolled in the study. Parental control will be applied for the pediatric population when needed.
13. Allergy, sensitivity or intolerance to concomitant drugs or excipients (Hypersensitivity to any of the excipients listed in section 6.1 or to bovine serum and murine 3T3-J2 cells);
14. Contraindications to the local or systemic antibiotics and/ or corticosteroids foreseen by the protocol;
15. Contraindications to the surgical procedure;
16. Clinically significant or unstable concurrent disease or other clinical contraindications to stem cell transplantation based upon investigator's judgment or other concomitant medical conditions affecting grafting procedure;
17. Patients (or parents in case of paediatric subject) unlikely to comply with the study protocol or unable to understand the nature and scope of the study or the possible benefits or unwanted effects of the study procedures and treatments.
18. Participation in another clinical trial where investigational drug was received less than 4 weeks prior to screening visit.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2015-10 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Success of transplantation | 12 months after transplantation
  The percentage of patients with a success of first transplantation at approximately 12 months from the first Holoclar treatment. Transplantation success is defined on the basis of the degree of "superficial corneal neo-vascularization" (CNV) and "epithelial defects".

SECONDARY OUTCOMES:
Success of one or two transplantation(s) | 12 months after the last transplantation
  The percentage of patients with clinical success after one or two ACLSCTs assessed at 12 months after the last treatment with Holoclar.
  Transplantation will be considered successful on the basis of the degree of "superficial corneal neo-vascularization" and "epithelial defects" according to the same definition as for the primary efficacy endpoint assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Graziella Pellegrini, Professor, Study Director — Holostem s.r.l.; Paolo Rama, MD, Principal Investigator — Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) Ospedale San Raffaele
Locations (1):
- Hospital San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No